CLINICAL TRIAL: NCT07361900
Title: Comparative Analysis of Botox, Occlusal Splints and Traditional Management of Bruxism in Patients With Implant Overdenture: A Randomized Controlled Trial.
Brief Title: Management of Bruxism in Patients With Implant Overdenture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Wafaa Ibrahim, Associate Professor, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FODMRC-2024-00100
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bruxism
Keywords: implant overdenture; Botox; Bruxism; Splint
MeSH Terms: conditions — Bruxism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botox injection (Active Comparator): Botox Administration Botulinum toxin type A (BTX-A; Botox, Allergan, Inc., Irvine, CA, USA) was administered through intramuscular injection into the masseter and temporalis muscles during a single treatment session. The masseter muscle received 30 units of BTX-A, while the temporalis muscle received 25 units. All injections were guided by electromyography
  Interventions: Drug: Botulinium toxin type A injection
- Maxillary Occlusal Stabilization Splint (Active Comparator): A maxillary full-arch hard clear acrylic muscle stabilization splint was fabricated for each participant. Each splint underwent intraoral evaluation to ensure optimal fit, retention, and stability on the maxillary dentition.
  Interventions: Device: Maxillary Occlusal Stabilization Splint
- Removal of overdenture (No Intervention): Overdentures were removed at night

INTERVENTIONS:
Drug: Botulinium toxin type A injection — Botulinum toxin type A (BTX-A; Botox, Allergan, Inc., Irvine, CA, USA) was administered through intramuscular injection into the masseter and temporalis muscles during a single treatment session. The masseter muscle received 30 units of BTX-A, while the temporalis muscle received 25 units. All injections were guided by electromyography (EMG).
  Other Names: Botox
  Arms: Botox injection
Device: Maxillary Occlusal Stabilization Splint — A maxillary full-arch hard clear acrylic muscle stabilization splint was fabricated for each participant
  Arms: Maxillary Occlusal Stabilization Splint

SUMMARY:
Objective To compare the effects of botulinum toxin type A (BTX-A) injections, occlusal stabilization splint therapy, and nocturnal overdenture removal on masticatory muscle activity and overdenture retention in patients with sleep bruxism wearing implant-retained mandibular overdentures.

Methods This randomized, single-blind, parallel-group clinical trial allocated patients with definite sleep bruxism to one of three groups (1:1:1): BTX-A injections with nocturnal overdenture wear, occlusal stabilization splint therapy with nocturnal overdenture wear, or nocturnal overdenture removal (control). Electromyographic (EMG) activity of the masseter and temporalis muscles was assessed at baseline and at 3, 6, 9, and 12 months. Overdenture retention was measured at 1, 3, 6, and 12 months using a digital force gauge. Intergroup comparisons were performed using one-way ANOVA with Tukey's post hoc test, and intragroup comparisons using repeated-measures ANOVA (α = 0.05).

DETAILED DESCRIPTION:
Diagnosis of sleep bruxism Electromyography (EMG) is a valuable tool for diagnosing sleep bruxism (SB), as it records electrical activity in the masticatory muscles (e.g., masseter and temporalis) during sleep, providing objective data on the frequency, duration, and intensity of muscle contractions. Unlike subjective patient reports or clinical examinations, EMG can detect SB episodes even when patients are unaware of their bruxism, which occurs in up to 80% of cases. While polysomnography (PSG) remains the gold standard for SB diagnosis due to its comprehensive monitoring of brain activity, muscle movements, and other physiological parameters, ambulatory EMG offers a more practical and accessible alternative for clinical settings. Despite this, EMG is widely used in research and clinical practice, particularly when combined with patient history and clinical examination, to achieve a reliable SB diagnosis conducted the assessments to minimize measurement bias.

Prosthetic Protocol

All participants received newly fabricated ODs to replace existing prostheses with compromised artificial dentition. The prosthetic rehabilitation included:

1. Installation of medium-retention nylon caps within metal housings to ensure consistent retention parameters
2. Restoration of opposing partially edentulous arches with fixed partial dentures
3. A one-month adaptation period incorporating necessary occlusal adjustments and prosthetic modifications Intervention Protocols Throughout the study duration, distinct wearing protocols were implemented for each experimental group: Groups I and II maintained continuous OD wear during sleep. Group I received BTX-A injection; Group II received additional intervention through conventional maxillary occlusal stabilization splints and Group III (Control Group) participants were instructed to remove their overdentures (ODs) during nocturnal sleep periods.

Group I protocol:

Botox Administration Botulinum toxin type A (BTX-A; Botox, Allergan, Inc., Irvine, CA, USA) was administered through intramuscular injection into the masseter and temporalis muscles during a single treatment session. The masseter muscle received 30 units of BTX-A, while the temporalis muscle received 25 units. All injections were guided by electromyography (EMG).

Reconstitution of BTX-A BTX-A reconstitution and syringe preparation were performed on a plastic-lined paper towel. The lyophilized BTX-A was reconstituted with 0.9% sodium chloride (normal saline) to achieve a final concentration of 10 units/0.1 mL. The precise volume of diluent, as outlined in the product insert, was drawn into a reconstitution syringe. The needle was then carefully inserted into the vial, which was positioned at a 45° angle. Saline was gently injected towards the vial walls to prevent BTX-A denaturation from bubbling or vigorous agitation. The presence of a vacuum within the vial confirmed its sterility. The vacuum was released by detaching the syringe from the needle, allowing atmospheric air to enter the vial. The reconstituted solution was visually inspected for clarity and the absence of particulate matter, appearing as a clear, colorless to slightly yellow solution. The solution was then drawn into the injection syringe by positioning the needle at the vial's bottom corner for complete extraction, after which the syringe was disconnected from the vial.

BTX-A Injection Protocol The reconstituted BTX-A solution was utilized immediately after preparation. Patients were seated in a comfortable upright position without head support, ensuring the Frankfort horizontal plane was parallel to the floor. No topical, local, or general anesthesia was administered prior to or during the injection procedure. The injection site on the patient's skin was disinfected using povidone-iodine U.S.P. 10% W/V.

A hollow, Teflon-coated, monopolar, disposable 27-gauge, 37-mm hypodermic needle electrode was employed for both muscle localization and drug delivery. This electrode was connected via a specialized cable to an audio-amplified electromyographic apparatus. A reference electrode was positioned centrally on the patient's forehead, with conductivity enhanced by applying conductive paste after thorough skin cleaning with alcohol. A ground electrode was placed on the forearm.

For the masseter muscle, anatomical landmarks were identified by palpation during clenching. Accurate needle tip placement was confirmed by a discernible "pop" upon fascial plane penetration, followed by positive EMG activity during clenching and the absence of EMG activity at rest. The EMG apparatus provided both auditory and visual feedback of muscle activity. For the temporalis muscle, the hypodermic needle electrode was inserted into the muscle fibers posterior to the frontal process of the zygomatic bone, approximately 1.5 to 2 cm superior to the zygomatic arch.

Upon proper needle positioning, aspiration was performed to confirm that the needle tip was not within a blood vessel. The reconstituted BTX-A was then injected slowly and gently after instructing the patient to relax the muscle. Post-injection, patients were advised to avoid strenuous physical activity for 24 hours, refrain from lying down for four to five hours following treatment, and to avoid massaging the treated area. Patients were also instructed to report BTX-A injections as part of their medical history. The procedure was repeated every 6 months for one year. All procedures were carried out by a certified practitioner (SM) throughout the study.

Group II Specific Protocol:

Maxillary Occlusal Stabilization Splint A maxillary full-arch hard clear acrylic muscle stabilization splint was fabricated for each participant in Group II. Each splint underwent intraoral evaluation to ensure optimal fit, retention, and stability on the maxillary dentition. Occlusal adjustments and refinements were meticulously performed directly in the patient's mouth. Following occlusal refinement, the splint was meticulously smoothed and polished to prevent irritation to adjacent soft tissues. Comprehensive instructions regarding splint usage and maintenance were provided to each patient. Compliance with nightly wear was required for the entire 12-month study period.

Electromyographic Analysis Protocol Patients' muscle activity was evaluated at baseline (one month from new overdenture insertion), and at 3, 6,9, and 12 months using electromyographic quantitative interference pattern analysis (QIPA) QIPA was conducted through surface EMG recordings of masseter and temporalis muscle activity during maximal voluntary clenching. The acquisition parameters were standardized as follows: Sweep speed: 100 ms/division, Sensitivity: 1 mV/division, and Bandpass filter: 20 Hz to 10 kHz.

The interference pattern analysis evaluated three key parameters:

1. Mean amplitude (mV): Calculated as the average potential difference between successive turns
2. Turn count: Quantified as the number of potential reversals exceeding 100 μV/ms, irrespective of baseline
3. Activity percentage: Representing the density of electromyographic activity within the interference pattern For each muscle group (masseter and temporalis), twenty consecutive recordings were obtained and analyzed to ensure data reliability.

The surface electrodes were positioned on the superficial masseter and anterior temporalis muscle and these positions were transferred to the clear template which was pierced at these points. Alcohol swabs (70% isopropyl alcohol) were used to clean their skin at the marked positions. The ground electrode was positioned on the forehead. Conductive EEG paste was filled on the inner sides of the electrodes. Adhesive tape was used to fix the reference electrodes on the corresponding positions. During silent reading by the patients, the right and left temporalis and masseter muscle's surface EMG activity was recorded.

All EMG'S tests were performed for all patients by the same assessor and under the same environmental conditions. The technique used and the guidelines were previously explained to the patient.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of definite sleep bruxism (SB)
* retention of natural dentition in the maxillary dental arch, without missing a single tooth of 6 anterior teeth, with no more than one or two missing premolar or molar teeth per quadrant
* existing implant-retained single overdentures (OD) that had been functionally loaded for at least one year prior to study initiation

Exclusion Criteria:

* had undergone any previous therapeutic interventions for bruxism
* exhibited medical conditions with known impacts on temporomandibular joint (TMJ) function, including (but not restricted to) post-radiation effects, osteoarthritis, or trauma-related pathologies.
* Any contraindication for BTX-A injection such as, allergy, pregnancy, and lactation.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Retention | 1month, 3 months, 6 months, 12 months
  For all groups, retention of the implant-supported overdenture was measured using a digital force gauge device

SECONDARY OUTCOMES:
II. Electromyography | 1 months, 3 months, 6 months, 12 months
  Patients' muscle activity was evaluated at baseline using electromyographic quantitative interference pattern analysis (QIPA). QIPA was conducted through surface EMG recordings of masseter and temporalis muscle activity during maximal voluntary clenching.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa I Ibrahim, Assoc. Prof., Principal Investigator — Associate Professor
Locations (1):
- Delta University for Science and Technology, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No